CLINICAL TRIAL: NCT05442008
Title: Study of Early MIDAS Reduction at 3 Months as Predictor of Long-term Erenumab Treatment in Chronic Migraine: a Real-life, Open-label, Trial
Brief Title: Predictive Role of MIDAS Reduction at 3 Months for Erenumab Treatment
Acronym: Ere-MIDAS
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ERENUMAB2022
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Migraine
Keywords: Migraine; Headache; CGRP; Monoclonal antibodies; Pain; Chronic migraine
MeSH Terms: conditions — Migraine Disorders; Headache; Pain | interventions — erenumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Erenumab 70/140 mg s.c. — Monoclonal antibody directed against the receptor of the Calcitonin Gene Related Peptide (CGRP)

SUMMARY:
In 2021, the Italian Medicines Agency approved reimbursement of monoclonal antibodies targeting the CGRP pathway (CGRP-mAbs) as preventive therapies for patients with high frequency and chronic migraine (CM). A moderate to severe disability, quantified as a MIgraine Disability ASsessment (MIDAS) score > or equal to 11, is required for prescription. Score reduction of at least 50% after the first three months (T3) is mandatory to continue treatment.

This is a prospective real-life, open-label study. CM patients will be treated with erenumab 70-140 mg subcutaneous injections every 28 days for one year (T13). We will record the following parameters: demographic and headache features, monthly migraine and headache days (MMDs and MHDs respectively), days and doses of symptomatic intake. Patients also completed questionnaires evaluating migraine related disability (MIDAS and HIT-6), psychological comorbidities (HADS-A and HADS-D), quality of life (MSQ and 0 to 100 visual analogue scale) and allodynia (ASC-12).

At least a 50% reduction in MIDAS score or MMDs after 3 months of treatment will be testedas predictors of long-term clinical outcome.

DETAILED DESCRIPTION:
Monoclonal antibodies directed against the Calcitonin Gene Related Peptide (CGRP-mAbs) pathway are a silver lining in the setting of migraine therapies, partly overcoming the issues related to poor effectiveness and tolerability of previous preventive treatments.

These drugs act on the CGRP pathway, a key vasoactive neuropeptide in migraine pathophysiology involved in activation and sensitization of afferent trigeminal nociceptors of the trigeminovascular system. Galcanezumab, fremanezumab and eptinezumab target the CGRP ligand, while erenumab, a fully human IgG2, targets its receptor. mAbs efficacy and safety have been largely documented in multiple randomized clinical trials, open-label studies as well as in the real-world setting.

The Italian Medicines Agency (AIFA) approved a 12-month period of mAbs treatment reimbursement through the National Health Service for migraine patients with the following features: i) at least 8 migraine days per month in the last three months, ii) a MIgraine Disability ASsessment (MIDAS) score ≥ 11, and iii) previous failure for inefficacy or no tolerability of at least three preventive drugs, among β-blockers, tricyclic antidepressants, antiepileptics, and onabotulinumtoxin-A for chronic migraine (CM).

In addition, a reduction of at least 50% of MIDAS score after 3 and 6 months of treatment is the only mandatory step to continue beyond these check-points. Thus, MIDAS score is pivotal for mAbs treatment initiation and continuation. MIDAS is a self-administered five-item questionnaire focusing on reduction in home and workplace productivity, and a score > 11 identify a set of patients with a moderate to severe disability. A MIDAS score reduction during mAbs treatment was demonstrated in the short and long term period, but its role as predictor of mAbs clinical outcome has never been consistently studied. A major concern for using a single parameter as a mandatory criterion for prescription and continuation of a preventive treatment is the limited ability to capture the multifaced disability that characterize the migraine spectrum. On the other side, reduction in monthly migraine days (MMDs) represents a pivotal outcome for clinical trials and physicians, but this may not completely highlight the patients' perspective.

The investigators consecutively screened migraine patients attending the outpatient clinic of the Headache Science & Neurorehabilitation Center of the IRCCS Mondino Foundation (Pavia, Italy).

The patients underwent a 1-year treatment with erenumab subcutaneous administration every 28 days (13 administrations) outside of the AIFA reimbursement program within a compassionate program.

During a baseline visit (T0), a neurologist with expertise in the headache field provided clinical indication to erenumab. At T0, the investigators checked the inclusion/exclusion criteria and the headache diaries of the three preceding months, and performed a full neurologic and general examination and a thorough anamnestic evaluation.

Patients who agreed to participate in the study signed a written informed consent and completed the baseline procedures, including clinical and demographic data recording and completion of a set of questionnaires to assess migraine related disability (MIDAS and HIT-6), psychological comorbidities (HADS-A and HADS-D), quality of life (MSQ), a self-perception of general health (0 to 100 visual analogue scale), and allodynia (ASC-12).

The first erenumab administration (70 mg) was delivered in the hospital setting at T0. After the first administration the patients were observed for 2 hours to monitor possible acute adverse events. The patients were then instructed to perform the following self-administrations of erenumab at home every 28 days (T1 to T12).

The patients returned to the Center every 12 weeks for the follow-up visits (T3 - T6 - T9 - T12), and at T13 for the last visit of the protocol. Monthly headache days (MHDs), monthly migraine days (MMDs), and days of acute drug intake were prospectively recorded in a paper headache diary. At each follow-up visit, the patients completed the same study procedures and clinical scales previously defined. At T3, erenumab dosage was increased in 72 patients up to 140 mg, according to the physician's judgment. All patients were allowed to keep their oral preventive medication with a stable dose across all study period.

The primary outcome was to evaluate the role of MIDAS reduction of at least 50% at T3 (MIDASRes) as a predictor of the long-term clinical outcome. As co-primary outcome, the investigators explored the role of early (T3) 50% MMDs reduction (MMDRes) as predictor of long-term efficacy.

In addition, the investigators evaluated the association between MIDASRes as well as MMDRes and the percentage of patients with a reduction in MMDs of at least 50% in the last 4 weeks of observation period (T13) when compared to baseline (RespondersT13). ResponderT13 were defined according to the IHS Guidelines for clinical trials involving CM patients.

As secondary outcomes, the investigators searched for possible associations between baseline clinical/demographic features and long-term efficacy of erenumab treatment, while, as exploratory outcomes, we described 1-year change in migraine-related disability, anxiety and depression severity, allodynia, and quality of life. The study was approved by the local Ethics Committee (P-20190105434).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CM according to ICHD-3 criteria for at least 12 months prior to enrollment;
* completion of a full headache diary in the 3 months preceding the enrollment; compliance to complete a daily headache diary for 1 year;
* previous failure of at least 3 classes of preventive treatments among beta-blockers, antiepileptic drugs, antidepressants, or onabotulinumtoxin-A;
* MIDAS score > 11.

Exclusion Criteria:

* severe cardiologic comorbidities;
* pregnancy and breastfeeding;
* previous adverse reaction to latex

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic migraine with clinical features in agreement with AIFA regulations for CGRP-mAbs prescription.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Predictive role of early MIDAS score reduction | Reduction in MMDs across 1-year treatment period
  To evaluate whether a >50% reduction in the MIDAS score at T3 (MIDAS-Res) is predictive of a more pronounced reduction in MMDs during a 1-year erenumab treatment.
Predictive role of early MMDs score reduction | Reduction in MMDs across 1-year treatment period
  To evaluate whether a >50% reduction in the monthly migraine days (MMDs) at T3 (MMD-Res) is predictive of a more pronounced reduction in MMDs during a 1-year erenumab treatment.

SECONDARY OUTCOMES:
Association between MIDAS-Res or MMD-Res and Responders at the end of the 1-year erenumab treatment | MIDAS-Res and MMD-Res defined after three months of erenumab treatment. ResponderT13 defined in the last 4 weeks of the 1-year erenumab treatment.
  Association between MIDAS-Res or MMD-Res and the percentage of patients with a reduction in MMDs of at least 50% in the last 4 weeks of observation period (T13) when compared to baseline (RespondersT13).

CONTACTS AND LOCATIONS:
Locations (1):
- Headache Science & Neurorehabilitation Center, Pavia, Italy

REFERENCES:
- [Background] Hepp Z, Dodick DW, Varon SF, Gillard P, Hansen RN, Devine EB. Adherence to oral migraine-preventive medications among patients with chronic migraine. Cephalalgia. 2015 May;35(6):478-88. doi: 10.1177/0333102414547138. Epub 2014 Aug 27. PMID 25164920
- [Background] Edvinsson L, Haanes KA, Warfvinge K, Krause DN. CGRP as the target of new migraine therapies - successful translation from bench to clinic. Nat Rev Neurol. 2018 Jun;14(6):338-350. doi: 10.1038/s41582-018-0003-1. PMID 29691490
- [Background] Scuteri D, Adornetto A, Rombola L, Naturale MD, Morrone LA, Bagetta G, Tonin P, Corasaniti MT. New Trends in Migraine Pharmacology: Targeting Calcitonin Gene-Related Peptide (CGRP) With Monoclonal Antibodies. Front Pharmacol. 2019 Apr 9;10:363. doi: 10.3389/fphar.2019.00363. eCollection 2019. PMID 31024319
- [Background] Tepper S, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein S, Winner P, Leonardi D, Mikol D, Lenz R. Safety and efficacy of erenumab for preventive treatment of chronic migraine: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017 Jun;16(6):425-434. doi: 10.1016/S1474-4422(17)30083-2. Epub 2017 Apr 28. PMID 28460892
- [Background] Barbanti P, Aurilia C, Egeo G, Fofi L, Cevoli S, Colombo B, Filippi M, Frediani F, Bono F, Grazzi L, Salerno A, Mercuri B, Carnevale A, Altamura C, Vernieri F. Erenumab in the prevention of high-frequency episodic and chronic migraine: Erenumab in Real Life in Italy (EARLY), the first Italian multicenter, prospective real-life study. Headache. 2021 Feb;61(2):363-372. doi: 10.1111/head.14032. Epub 2020 Dec 18. PMID 33337544
- [Background] Sacco S, Amin FM, Ashina M, Bendtsen L, Deligianni CI, Gil-Gouveia R, Katsarava Z, MaassenVanDenBrink A, Martelletti P, Mitsikostas DD, Ornello R, Reuter U, Sanchez-Del-Rio M, Sinclair AJ, Terwindt G, Uluduz D, Versijpt J, Lampl C. European Headache Federation guideline on the use of monoclonal antibodies targeting the calcitonin gene related peptide pathway for migraine prevention - 2022 update. J Headache Pain. 2022 Jun 11;23(1):67. doi: 10.1186/s10194-022-01431-x. PMID 35690723
- [Background] Stewart WF, Lipton RB, Kolodner KB, Sawyer J, Lee C, Liberman JN. Validity of the Migraine Disability Assessment (MIDAS) score in comparison to a diary-based measure in a population sample of migraine sufferers. Pain. 2000 Oct;88(1):41-52. doi: 10.1016/S0304-3959(00)00305-5. PMID 11098098
- [Background] Iannone LF, Fattori D, Benemei S, Chiarugi A, Geppetti P, De Cesaris F. Long-Term Effectiveness of Three Anti-CGRP Monoclonal Antibodies in Resistant Chronic Migraine Patients Based on the MIDAS score. CNS Drugs. 2022 Feb;36(2):191-202. doi: 10.1007/s40263-021-00893-y. Epub 2022 Feb 11. PMID 35146696
- [Background] Lipton RB, Tepper SJ, Reuter U, Silberstein S, Stewart WF, Nilsen J, Leonardi DK, Desai P, Cheng S, Mikol DD, Lenz R. Erenumab in chronic migraine: Patient-reported outcomes in a randomized double-blind study. Neurology. 2019 May 7;92(19):e2250-e2260. doi: 10.1212/WNL.0000000000007452. Epub 2019 Apr 17. PMID 30996060
- [Background] Ashina M, Goadsby PJ, Reuter U, Silberstein S, Dodick DW, Xue F, Zhang F, Paiva da Silva Lima G, Cheng S, Mikol DD. Long-term efficacy and safety of erenumab in migraine prevention: Results from a 5-year, open-label treatment phase of a randomized clinical trial. Eur J Neurol. 2021 May;28(5):1716-1725. doi: 10.1111/ene.14715. Epub 2021 Jan 20. PMID 33400330
- [Background] Goadsby PJ, Reuter U, Lanteri-Minet M, Paiva da Silva Lima G, Hours-Zesiger P, Fernandes C, Wen S, Tenenbaum N, Kataria A, Ferrari MD, Klatt J. Long-term Efficacy and Safety of Erenumab: Results From 64 Weeks of the LIBERTY Study. Neurology. 2021 May 31;96(22):e2724-e2735. doi: 10.1212/WNL.0000000000012029. PMID 33910942
- [Background] Tassorelli C, Diener HC, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of chronic migraine in adults. Cephalalgia. 2018 Apr;38(5):815-832. doi: 10.1177/0333102418758283. Epub 2018 Mar 4. PMID 29504482
- [Background] Alpuente A, Gallardo VJ, Caronna E, Torres-Ferrus M, Pozo-Rosich P. In search of a gold standard patient-reported outcome measure to use in the evaluation and treatment-decision making in migraine prevention. A real-world evidence study. J Headache Pain. 2021 Dec 13;22(1):151. doi: 10.1186/s10194-021-01366-9. PMID 34903177
- [Background] Iannone LF, Fattori D, Benemei S, Chiarugi A, Geppetti P, De Cesaris F. Predictors of sustained response and effects of the discontinuation of anti-calcitonin gene related peptide antibodies and reinitiation in resistant chronic migraine. Eur J Neurol. 2022 May;29(5):1505-1513. doi: 10.1111/ene.15260. Epub 2022 Feb 13. PMID 35098620
- [Background] Vernieri F, Brunelli N, Messina R, Costa CM, Colombo B, Torelli P, Quintana S, Cevoli S, Favoni V, d'Onofrio F, Egeo G, Rao R, Filippi M, Barbanti P, Altamura C. Discontinuing monoclonal antibodies targeting CGRP pathway after one-year treatment: an observational longitudinal cohort study. J Headache Pain. 2021 Dec 18;22(1):154. doi: 10.1186/s10194-021-01363-y. PMID 34922444
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] De Icco R, Fiamingo G, Greco R, Bottiroli S, Demartini C, Zanaboni AM, Allena M, Guaschino E, Martinelli D, Putorti A, Grillo V, Sances G, Tassorelli C. Neurophysiological and biomolecular effects of erenumab in chronic migraine: An open label study. Cephalalgia. 2020 Oct;40(12):1336-1345. doi: 10.1177/0333102420942230. Epub 2020 Jul 26. PMID 32715736
- [Background] Bottiroli S, De Icco R, Vaghi G, Pazzi S, Guaschino E, Allena M, Ghiotto N, Martinelli D, Tassorelli C, Sances G. Psychological predictors of negative treatment outcome with Erenumab in chronic migraine: data from an open label long-term prospective study. J Headache Pain. 2021 Oct 2;22(1):114. doi: 10.1186/s10194-021-01333-4. PMID 34600468
- [Background] Giannouchos TV, Mitsikostas DD, Ohsfeldt RL, Vozikis A, Koufopoulou P. Cost-Effectiveness Analysis of Erenumab Versus OnabotulinumtoxinA for Patients with Chronic Migraine Attacks in Greece. Clin Drug Investig. 2019 Oct;39(10):979-990. doi: 10.1007/s40261-019-00827-z. PMID 31302899
- [Background] Burch RC, Buse DC, Lipton RB. Migraine: Epidemiology, Burden, and Comorbidity. Neurol Clin. 2019 Nov;37(4):631-649. doi: 10.1016/j.ncl.2019.06.001. Epub 2019 Aug 27. PMID 31563224
- [Background] Berra E, Sances G, De Icco R, Avenali M, Berlangieri M, De Paoli I, Bolla M, Allena M, Ghiotto N, Guaschino E, Cristina S, Tassorelli C, Sandrini G, Nappi G. Cost of Chronic and Episodic Migraine. A pilot study from a tertiary headache centre in northern Italy. J Headache Pain. 2015;16:532. doi: 10.1186/s10194-015-0532-6. Epub 2015 May 27. PMID 26018292
- [Background] Tepper SJ, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein SD, Winner P, Zhang F, Cheng S, Mikol DD. Long-term safety and efficacy of erenumab in patients with chronic migraine: Results from a 52-week, open-label extension study. Cephalalgia. 2020 May;40(6):543-553. doi: 10.1177/0333102420912726. Epub 2020 Mar 26. PMID 32216456
- [Background] Barbanti P, Aurilia C, Cevoli S, Egeo G, Fofi L, Messina R, Salerno A, Torelli P, Albanese M, Carnevale A, Bono F, D'Amico D, Filippi M, Altamura C, Vernieri F; EARLY Study Group. Long-term (48 weeks) effectiveness, safety, and tolerability of erenumab in the prevention of high-frequency episodic and chronic migraine in a real world: Results of the EARLY 2 study. Headache. 2021 Oct;61(9):1351-1363. doi: 10.1111/head.14194. Epub 2021 Jul 26. PMID 34309862
- [Background] Becker WJ, Spacey S, Leroux E, Giammarco R, Gladstone J, Christie S, Akaberi A, Power GS, Minhas JK, Mancini J, Rochdi D, Filiz A, Bastien N. A real-world, observational study of erenumab for migraine prevention in Canadian patients. Headache. 2022 Apr;62(4):522-529. doi: 10.1111/head.14291. Epub 2022 Apr 10. PMID 35403223
- [Background] Lambru G, Hill B, Murphy M, Tylova I, Andreou AP. A prospective real-world analysis of erenumab in refractory chronic migraine. J Headache Pain. 2020 Jun 1;21(1):61. doi: 10.1186/s10194-020-01127-0. PMID 32487102
- [Background] Zecca C, Cargnin S, Schankin C, Giannantoni NM, Viana M, Maraffi I, Riccitelli GC, Sihabdeen S, Terrazzino S, Gobbi C. Clinic and genetic predictors in response to erenumab. Eur J Neurol. 2022 Apr;29(4):1209-1217. doi: 10.1111/ene.15236. Epub 2022 Jan 21. PMID 34965002
- [Background] Baraldi C, Castro FL, Cainazzo MM, Pani L, Guerzoni S. Predictors of response to erenumab after 12 months of treatment. Brain Behav. 2021 Aug;11(8):e2260. doi: 10.1002/brb3.2260. Epub 2021 Jul 16. PMID 34268907
- [Background] Silvestro M, Tessitore A, Scotto di Clemente F, Battista G, Tedeschi G, Russo A. Refractory migraine profile in CGRP-monoclonal antibodies scenario. Acta Neurol Scand. 2021 Sep;144(3):325-333. doi: 10.1111/ane.13472. Epub 2021 May 21. PMID 34019304
- [Background] Schoenen J, Timmermans G, Nonis R, Manise M, Fumal A, Gerard P. Erenumab for Migraine Prevention in a 1-Year Compassionate Use Program: Efficacy, Tolerability, and Differences Between Clinical Phenotypes. Front Neurol. 2021 Dec 10;12:805334. doi: 10.3389/fneur.2021.805334. eCollection 2021. PMID 34956071
- [Background] Vernieri F, Altamura C, Brunelli N, Costa CM, Aurilia C, Egeo G, Fofi L, Favoni V, Lovati C, Bertuzzo D, d'Onofrio F, Doretti A, Di Fiore P, Finocchi C, Schiano Di Cola F, Ranieri A, Colombo B, Bono F, Albanese M, Cevoli S, Barbanti P; GARLIT Study Group. Rapid response to galcanezumab and predictive factors in chronic migraine patients: A 3-month observational, longitudinal, cohort, multicenter, Italian real-life study. Eur J Neurol. 2022 Apr;29(4):1198-1208. doi: 10.1111/ene.15197. Epub 2021 Dec 6. PMID 34826192
- [Background] Vernieri F, Altamura C, Brunelli N, Costa CM, Aurilia C, Egeo G, Fofi L, Favoni V, Pierangeli G, Lovati C, Aguggia M, d'Onofrio F, Doretti A, Di Fiore P, Finocchi C, Rao R, Bono F, Ranieri A, Albanese M, Cevoli S, Barbanti P; GARLIT Study Group. Galcanezumab for the prevention of high frequency episodic and chronic migraine in real life in Italy: a multicenter prospective cohort study (the GARLIT study). J Headache Pain. 2021 May 3;22(1):35. doi: 10.1186/s10194-021-01247-1. PMID 33941080
- [Background] Ornello R, Baraldi C, Guerzoni S, Lambru G, Fuccaro M, Raffaelli B, Gendolla A, Barbanti P, Aurilia C, Cevoli S, Favoni V, Vernieri F, Altamura C, Russo A, Silvestro M, Dalla Valle E, Mancioli A, Ranieri A, Alfieri G, Latysheva N, Filatova E, Talbot J, Cheng S, Holle D, Scheffler A, Nezadal T, Ctrnacta D, Sipkova J, Matousova Z, Sette L, Casalena A, Maddestra M, Viola S, Affaitati G, Giamberardino MA, Pistoia F, Reuter U, Sacco S. Gender Differences in 3-Month Outcomes of Erenumab Treatment-Study on Efficacy and Safety of Treatment With Erenumab in Men. Front Neurol. 2021 Dec 16;12:774341. doi: 10.3389/fneur.2021.774341. eCollection 2021. PMID 34975732
- [Background] Sacco S, Braschinsky M, Ducros A, Lampl C, Little P, van den Brink AM, Pozo-Rosich P, Reuter U, de la Torre ER, Sanchez Del Rio M, Sinclair AJ, Katsarava Z, Martelletti P. European headache federation consensus on the definition of resistant and refractory migraine : Developed with the endorsement of the European Migraine & Headache Alliance (EMHA). J Headache Pain. 2020 Jun 16;21(1):76. doi: 10.1186/s10194-020-01130-5. PMID 32546227
- [Background] Ailani J, Burch RC, Robbins MS; Board of Directors of the American Headache Society. The American Headache Society Consensus Statement: Update on integrating new migraine treatments into clinical practice. Headache. 2021 Jul;61(7):1021-1039. doi: 10.1111/head.14153. Epub 2021 Jun 23. PMID 34160823
- [Background] Ishii R, Schwedt TJ, Dumkrieger G, Lalvani N, Craven A, Goadsby PJ, Lipton RB, Olesen J, Silberstein SD, Burish MJ, Dodick DW. Chronic versus episodic migraine: The 15-day threshold does not adequately reflect substantial differences in disability across the full spectrum of headache frequency. Headache. 2021 Jul;61(7):992-1003. doi: 10.1111/head.14154. Epub 2021 Jun 3. PMID 34081791
- [Derived] De Icco R, Vaghi G, Allena M, Ghiotto N, Guaschino E, Martinelli D, Ahmad L, Corrado M, Bighiani F, Tanganelli F, Bottiroli S, Cammarota F, Sances G, Tassorelli C. Does MIDAS reduction at 3 months predict the outcome of erenumab treatment? A real-world, open-label trial. J Headache Pain. 2022 Sep 17;23(1):123. doi: 10.1186/s10194-022-01480-2. PMID 36115947